CLINICAL TRIAL: NCT01312935
Title: A Phase 2 Proof of Concept Study of PMX-60056 for the Reversal of Heparin in Patients Undergoing Percutaneous Coronary Intervention (PCI)
Brief Title: Reversal of Heparin in Patients Undergoing Percutaneous Coronary Intervention (PCI)
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: PolyMedix decided to stop enrollment in both clinical trials due to observations of reductions in blood pressure.
Sponsor: PolyMedix, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PMX56-203
Record Dates: First submitted 2011-03-08; First posted 2011-03-11 (Estimated); Last update posted 2012-05-17 (Estimated); Status verified 2012-05

CONDITIONS: Percutaneous Coronary Intervention; Coronary Artery Disease (CAD); Angioplasty
Keywords: Percutaneous Coronary Intervention; Heparin; Angioplasty; LMWH
MeSH Terms: conditions — Coronary Artery Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Heparin and PMX-60056 (Experimental)
  Interventions: Drug: PMX-60056

INTERVENTIONS:
Drug: PMX-60056 — investigational drug

SUMMARY:
The study investigates the safety and efficacy of PMX-60056 for the Reversal of Heparin in Patients Undergoing Percutaneous Coronary Intervention (PCI)

DETAILED DESCRIPTION:
PMX-60056 is being developed as a rapid and effective reversal agent for use in those situations where anticoagulation by heparin, or LMWH must be quickly stopped. Potential uses include reversal of anticoagulation induced to prevent clotting during surgical procedures, and rescue from cases of inadvertent or unexpected overdose.

ELIGIBILITY:
Inclusion Criteria:

1. The patient will undergo PCI for diagnostic and/or therapeutic purposes with a procedure that uses anticoagulation before the instrumentation and reversal of anticoagulation immediately after the procedure.
2. Male or female patients of any race, aged 18-80 years old.
3. The patient will be anti-coagulated with unfractionated heparin.
4. The patient is medically stable and physically and mentally able to participate in this study.
5. The patient has given written informed consent to participate in this study after fully understanding the implications and constraints of the protocol.

Exclusion Criteria:

1. The patient requires emergency surgery under conditions which prevent compliance with this protocol or which might cause unacceptable risk to the patient.
2. The patient requires any concomitant surgical procedures (e.g., carotid artery, CABG) during the PCI.
3. The patient has received any investigational drug within 30 days of study enrollment, or has had any prior exposure to PMX-60056.
4. The patient has any condition or abnormality which may, in the opinion of the Investigator, compromise the safety of the patient.
5. The patient is pregnant or breast feeding.
6. The patient is of childbearing potential and not under adequate contraceptive protection.
7. The patient has a history of clinically significant hematologic disease including heparin-induced thrombocytopenia, bleeding disorders, or platelet count <100,000.
8. Severe impaired hepatic function (SGOT, SGPT >2 x ULN).
9. History of AIDS, ± HIV.
10. History of allergy to heparin (beef or pig), protamine, or salmon.
11. History of chronic alcohol or drug abuse within the last one year.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2011-04; Primary Completion 2012-06 (Estimated); Study Completion 2012-08 (Estimated)

PRIMARY OUTCOMES:
The primary outcome measure of this study is the ability to reverse the anticoagulant effects of heparin (as measured by ACT) to the same extent as is known for protamine. intravenous infusion of PMX-60056. | Immediately post completion of PCI procedure, until 2 hours after last dose.

CONTACTS AND LOCATIONS:
Locations (3):
- United States (3):
  - South Bend, Indiana
  - Detroit, Michigan
  - Rapid City, South Dakota